CLINICAL TRIAL: NCT03997682
Title: Hands-Up Program: Protocol for a Feasibility Study of a Combined Exercise and Education Randomized Controlled Trial of a 6-week Intervention in People With a Distal Radius Fracture
Brief Title: Hands-Up: Exercise and Education Program After a Wrist Fracture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Western University, Canada (Other)
Responsible Party: Principal Investigator, Joy MacDermid, Professor, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 114095
Record Dates: First submitted 2019-06-10; First posted 2019-06-25 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Distal Radius Fracture; Osteoporosis
MeSH Terms: conditions — Wrist Fractures; Osteoporosis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hands-Up Program (Experimental): Participants will be guided through a 45 minutes exercise program, set up as a group exercise class, with program modifications being made for each individual participant. In order to meet the requisite number of participants there will be approximately 4 cohorts of 10 participants. Immediately after the exercise class participants will attend a 30-minute educational session. The educational sessions will cover bone health principles, nutrition for bone health, osteoporosis practice guidelines, ways to self-monitor balance and lower extremity strength, impacts of physical activity, home hazard detection, hazards at work and in the community, postural effects on bone loading and fracture risk, and integrating physical activity in daily life. Nutritional education will emphasize the importance of calcium and vitamin D, sources of both diary and dairy free calcium, vitamin D supplements, the importance of protein, and meat and meat-free sources of protein.
  Interventions: Other: Hands-Up Program
- Standard Care (No Intervention): The control group will receive usual care after a distal radius fracture. The standard care for a distal radius fracture will receive an assessment related to whether casting or surgery is necessary. The participant may be in a cast for 6 weeks with routine check up and x-rays to monitor the healing, at 3 months, 6 months and 12 months. The participant should receive some physical therapy related to restoring function of the hand and wrist.

INTERVENTIONS:
Other: Hands-Up Program — In addition to the usual care, being allocated to the intervention group would require the participant to attend an exercise and education program once their cast has been removed and they've restored some strength and function in their hand and wrist. The exercise portion of the intervention will focus on strength and balance training, with aspects of managing our distal radius fracture healing as well. The education will focus on learning about risk factors for a distal radius fracture, osteoporosis, exercise for adults, nutrition for adults and falls prevention strategies.
  Arms: Hands-Up Program

SUMMARY:
Osteoporosis is a bone disease that increases the risk of fractures. People aged 50-65 diagnosed with osteoporosis feel too young to have the disease. But this happens. They need to learn how to modify their lifestyle to minimize the chances of fractures. In this age group, a wrist fracture is usually the first sign of osteoporosis. Fracture risk increases if they are not taught to exercise, eat properly, and identifies fall risk factors early in their diagnosis. Some studies have looked at interventions for osteoporosis in women over the age of 65, but by this age they have likely already had a spine fracture. No studies have addressed the early-onset osteoporosis age group, intervening before spine fractures occur. I will develop an exercise, nutrition, and falls prevention education program to improve the strength, balance and knowledge of people aged 50-65 who had an osteoporotic wrist fracture. I will use this treatment approach and determine if it is more effective than the usual way of treating people with wrist fractures, determining if this is a better strategy for managing osteoporosis. I will have two groups of patients. First, those, over six weeks, receive twice weekly classes that include exercise and education. Here the focus is on bone health and fracture prevention. The control will receive usual physical therapy and the educational materials at the end of their study participation. The treatment will be randomly allocated to 74 men and women between the ages of 50-65 years of age who are 6-10 weeks post-fracture. The outcomes on both groups will be assessed and compared. I will focus on hand function, balance, fall hazard detection, and a bone health behaviour checklist. Using these outcomes, I can determine which treatment approach works best. Osteoporosis affects one in three women and one in five men, making this an important study to improve the lives for many Canadians. The risk of osteoporosis fractures increases with age, making early interventions critical.

DETAILED DESCRIPTION:
Participants included in this study will be recruited from the Hand and Upper Limb Clinic (HULC) at St. Joseph's Hospital. Patients at HULC are routinely tested function and strength and use questionnaires that ask about pain and disability. These procedure help to monitor usual recovery. Participation in this study will require being screened for eligibility and informed about the study by their surgeon or their delegate,who is a research assistant working on this project. By using a computer-generated sequence, the participant will be randomly allocated to either of the following treatment groups:

1. Usual physical therapy OR
2. Usual physical therapy AND Hands-Up Program (Exercise and Education) The standard care for a distal radius fracture would include receiving an assessment related to whether casting or surgery is necessary. The participant may be in a cast for 6 weeks with routine check up and x-rays to monitor the healing, at 3 months, 6 months and 12 months. The participant should receive some physical therapy related to restoring function of the hand and wrist.

In addition to the usual care, being allocated to the intervention group would require the participant to attend an exercise and education program once their cast has been removed and they've restored some strength and function in their hand and wrist. The exercise portion of the intervention will focus on strength and balance training, with aspects of managing distal radius fracture healing as well. The education will focus on learning about risk factors for a distal radius fracture, osteoporosis, exercise for adults, nutrition for adults and falls prevention strategies. Both the exercise and education programs will take place at the HULC clinical research lab. The participant will be asked to come in two times per week for approximately 75 minutes per session. The participant will have 45 minutes of exercise which will include upper and lower body strength training, balance and some hand and wrist rehabilitation, followed by 30 minutes of education related to distal radius fractures, osteoporosis education, exercise, nutrition and falls prevention.

The control group will receive the educational materials (one-page info graphics) at the end of the 12-month study participation.

On the participant's initial visit, they will be asked to fill out questionnaires to assess their symptoms related with pain, disability and function. The investigators will conduct several strength assessments such as, a pinch strength test, grip strength, lower body strength and upper body strength. The investigators will take a bone mineral density assessment using a dual energy x-ray absorptiometry (DXA), of the spine, hip and wrist. Follow-up visits for the study will be similar to our usual follow-up, which takes place at 6 week, 3 month, 6 months and 12 months after the participant's initial visit. Specifically, at baseline the participant will be asked to have a DXA (an X-ray measuring your bone density), complete some questionnaires and perform strength and balance assessments. The DXA assessment will not be done at the 6 week, 3 month assessment, but the questionnaires and strength and balance assessments wee be done at those time points. At the 12 month mark all of the outcome assessments will be repeated, including the DXA. Additionally, a physical activity diary will be provided at the initial visit which will be maintained as a daily log of exercise and physical activity during the study period (for one-year). The participant will be asked to bring the physical activity diary to the follow-up visits (at 6 weeks, 3 months, 6 months, and 12 months) so that research staff can keep a copy of physical activity log completed during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Patient attending the Roth | McFarlane Hand and Upper Limb Clinic (HULC)
* Patients that have had a low-impact distal radius fracture (DRF) within the last 6-10 weeks
* Aged 50-65
* Able to speak and understand English
* Are able to provide informed consent

Exclusion Criteria:

* Any contraindications to exercise
* Progressive neurological disorders that would affect study participation
* Unable to stand or walk independently
* Unable to provide consent

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2021-03-10 (Estimated); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of recruitment | 12 months
  Number of participants recruited in one year. Recruitment will be feasible if 74 participants are recruited within 12 months
Feasibility of Retention | 12 months
  number of participants that attend the final study visit. Feasibility will be met if 75% of participants attend the final study visit.
Feasibility of Adherence | 12 months
  Number of participants attending each exercise class. Feasibility will be met if the participant attends greater than 60% of the exercise classes

SECONDARY OUTCOMES:
Grip Strength | 12 months
  Grip strength measured in kilograms using a grip strength dynamometer: Saehan, Saehan Corp. Masan, Korea.
Patient Rated Wrist Evaluation | 12 months
  Self-reported pain and function from the patient rated wrist evaluation. The overall score will be assessed at each time point. The overall score is out of 100. Units on a scale.
Bone Density | 12 months
  A t-score as measured by the DXA.
Osteoporosis Knowledge | 12 months
  An osteoporosis knowledge test, using a scale, out of 30.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Joseph Health Care, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
The individual participant data will not be made publicly available. Only de-identified data will be shared.

REFERENCES:
- [Derived] Ziebart C, MacDermid J, Bryant D, Szekeres M, Suh N. Hands-Up program: protocol for a feasibility randomised controlled trial of a combined 6-week exercise and education intervention in adults aged 50-65 with a distal radius fracture. BMJ Open. 2021 Jul 30;11(7):e046122. doi: 10.1136/bmjopen-2020-046122. PMID 34330854